CLINICAL TRIAL: NCT03908749
Title: A Real-world Clinical Study of Pyrotinib Maleate Tablets in the Treatment of Breast Cancer Patients With Positive Her-2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Yue-Yin Pan, Director, Anhui Provincial Hospital
Other Study IDs: AnhuiPH
Record Dates: First submitted 2019-04-07; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: HER2 Positive Breast Carcinoma
Keywords: Pyrotinib Maleate Tablets; HER-2; Real word study; Efficacy; Safety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the efficacy and safety of Pyrotinib Maleate Tablets in the treatment of advanced breast cancer patients with positive her-2.

DETAILED DESCRIPTION:
This study intends to carry out multicenter, observational cohort clinical research, using maleic acid pyrrole for his piece of HER-2 positive treatment of advanced breast cancer treatment, observation and verification maleic acid pyrrole for his piece for a line or a single drug resistance by bead in the real diagnosis and treatment in patients with advanced breast cancer environment and the efficacy and safety of new treatments. Biomarkers of breast cancer prognosis are of great significance in predicting the degree of malignancy, metastasis and recurrence of breast cancer, as well as guiding clinical treatment programs.This study will explore the prognostic factors and curative effect of breast cancer patients from multiple aspects, explore the dominant population of breast cancer patients with pyrrolidone maleate, and provide the theoretical basis for individualized treatment for clinical treatment practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients .
2. Confirmed by pathological examination of breast cancer patients with positive her-2 expression
3. The researchers determined that the standard neoadjuvant regimen was ineffective in the treatment of patients with locally advanced her-2 positive breast cancer or that the standard neoadjuvant regimen was not applicable.
4. Patients should be voluntary to the trial and provide with signed informed consent
5. The researchers believe patients can benefit from the study.

Exclusion Criteria:

1. Patients with a known history of allergic reactions and/or hypersensitivity attributed to Pyrotinib maleate tablets or its accessories
2. Pregnant or lactating women
3. Patients with Pyrotinib maleate tablets contraindications
4. Patients of doctors considered unsuitable for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced her-2 positive breast cancer who are not treated with standard neoadjuvant regimens or who are not treated with standard neoadjuvant regimens.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-10 (Estimated); Primary Completion 2020-04-10 (Estimated); Study Completion 2020-10-10 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  Progress free survival is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.
pCR | 1 year
  Pathological complete response is the breast primary focus and axillary lymph node surgery specimen pathological examination without invasive tumor cell residual

SECONDARY OUTCOMES:
OS | 1 year
  overall survival is defined as the length of time from random assignment to death or to last contact.
AE | 1 year
  adverse events are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.
ORR | 1 year
  Objective tumor response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments
DCR | 1 year
  Disease control rate (DCR) refers to the percentage of cases with remission and disease stability after treatment in the total number of evaluable cases
DFS | 1 year
  Disease-free survival (DFS) is defined as the time from the beginning of randomization to recurrence or death due to Disease progression
DDFS | 1 year
  Disease /recurrence free survival (DDFS) refers to a period of time after treatment for a tumor patient where no metastatic lesions were found anywhere else in the body except for the accident of the primary lesion

IPD SHARING:
Plan to Share IPD: Undecided